CLINICAL TRIAL: NCT02342574
Title: F901318 - A Phase I, Double-Blind, Placebo Controlled, Single and Multiple Ascending Intravenous Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Male Subjects
Brief Title: F901318 Multiple Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F901318-01-02-14
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-08

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — olorofim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (18):
- A active (Experimental): Six subjects receiving F901318 1.5 mg/kg intravenously for eight days
  Interventions: Drug: F901318
- A placebo (Placebo Comparator): Two subjects receiving F901318 placebo intravenously for eight days
  Interventions: Drug: Placebo
- B active (Experimental): Six subjects receiving F901318 3 mg/kg intravenously for eight days
  Interventions: Drug: F901318
- B placebo (Placebo Comparator): Two subjects receiving F901318 placebo intravenously for eight days
  Interventions: Drug: Placebo
- C active (Experimental): Six subjects receiving F901318 4 mg/kg intravenously for eight days
  Interventions: Drug: F901318
- C placebo (Placebo Comparator): Two subjects receiving F901318 placebo intravenously for eight days
  Interventions: Drug: Placebo
- D1 active (Experimental): Six subjects dosed for one day with F901318 intravenously dose to be determined
  Interventions: Drug: F901318
- D1 placebo (Placebo Comparator): Two subjects receiving F901318 placebo intravenously for one day
  Interventions: Drug: Placebo
- E1 active (Experimental): Six subjects dosed for one day with F901318 intravenously dose to be determined
  Interventions: Drug: F901318
- E1 placebo (Placebo Comparator): Two subjects receiving F901318 placebo intravenously for one day
  Interventions: Drug: Placebo
- F1 active (Experimental): Six subjects dosed for one day with F901318 intravenously dose to be determined
  Interventions: Drug: F901318
- F1 placebo (Placebo Comparator): Two subjects receiving F901318 placebo intravenously for one day
  Interventions: Drug: Placebo
- D2 active (Experimental): Six subjects dosed for eight days with F901318 intravenously dose to be determined
  Interventions: Drug: F901318
- D2 placebo (Placebo Comparator): Two subjects receiving F901318 placebo intravenously for eight days
  Interventions: Drug: Placebo
- E2 active (Experimental): Six subjects dosed for eight days with F901318 intravenously dose to be determined
  Interventions: Drug: F901318
- E2 placebo (Placebo Comparator): Two subjects receiving F901318 placebo intravenously for eight days
  Interventions: Drug: Placebo
- F2 active (Experimental): Six subjects dosed for eight days with F901318 intravenously dose to be determined
  Interventions: Drug: F901318
- F2 placebo (Placebo Comparator): Two subjects receiving F901318 placebo intravenously for eight days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: F901318 — Administration of active compound
  Arms: A active; B active; C active; D1 active; D2 active; E1 active; E2 active; F1 active; F2 active
Drug: Placebo — Administration of placebo
  Arms: A placebo; B placebo; C placebo; D1 placebo; D2 placebo; E1 placebo; E2 placebo; F1 placebo; F2 placebo

SUMMARY:
Double blind, placebo controlled, parallel group ascending dose study evaluating single and multiple (x8 days) dose levels of F901318 in groups of male healthy subjects with the objective of defining a dosing schedule for phase ll clinical trials. F901318, a novel and potent antifungal agent for the treatment of invasive aspergillosis, will be delivered intravenously in a range of dosing schedules driven by pharmacokinetic evaluation in real time. Safety and tolerability of those schedules will also be assessed.

DETAILED DESCRIPTION:
Double blind, placebo controlled, ascending single and multiple intravenous dose, sequential group study. This will be a study in two parts. In the first part, up to twenty four subjects will complete the study in up to 3 cohorts (Groups A to C), each group consisting of 8 subjects, six of whom will receive active compound and two will receive placebo for eight days. Each subject will be on study for approximately 7 weeks. Each subject will participate in one treatment cohort only, residing at the Clinical Research Unit (CRU) from Day -1 (the day before dosing) to Day 13 (120 hours post the last dose).

This first part (Part 1) will test doses already evaluated in the previous single ascending dose study (F901318-01-01-14, 0.25-4 mg/kg given over 4 hours). The dose levels for the study are expected to be 1.5, 3 and 4 mg/kg/day given as a four hour infusion once daily.

In the second part of the study (Part 2), doses higher than those previously evaluated may be studied and/or different dosing schedules designed to deliver a maximum tolerated dose over 24 hours. If a dose level higher than those previously studied is chosen, there will be an optional single dose studied initially for safety and pharmacokinetic profile (Part 2A), followed about 14 days later in another group of subjects by exposure at that same dose level over 8 consecutive days (Part 2B). These higher doses may be given in a once or twice daily dosing schedule. Six subjects will receive active compound and two will receive placebo in both the single dose and multiple dose cohorts. The single dose cohorts will receive study drug in a sentinel group design in which two subjects receive study drug (one active and one placebo) on the first day and the rest of the group one day later. There will be a review of safety data by the Principal Investigator and the Medical Monitor after the first two subjects have been dosed and before the last six subjects are dosed in each cohort in part 2A.

In Part 2, up to forty-eight subjects will complete the study in up to 6 cohorts (Part 2A, Groups D1 to F1, single day dosing, and Part 2B, Groups D2 to F2 eight days' dosing). Subjects in Parts 1 and 2B will be on the study for approximately 7 weeks and Part 2A for approximately 8 weeks. Each subject will participate in one treatment cohort only, residing at the Clinical Research Unit (CRU) from Day -1 (the day before dosing) to Day 6 (120 hours after the single dose in Parts 1 and 2A) and from Day -1 (the day before dosing) to Day 13 (120 hours after the first dose in Part 2B). The proposed total daily dose levels for Part 2 will be up to 10 mg/kg/day given either once daily or in two split daily doses. The duration of the infusions will be between 2 and 24 hours which may include a loading dose to achieve therapeutic plasma concentrations as quickly as possible.

All subjects will return for a post-study visit 8 to 10 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males of any ethnic origin between 18 and 45 years of age and weighing 60-100 kg inclusive
2. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is acceptable)
3. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions
4. Subjects must have ophthalmology assessments within the normal limits at screening. This includes normal Meibomian gland function

Exclusion Criteria:

1. Male subjects who are not willing to use appropriate contraception (such as a condom) during the study and until follow up
2. Subjects who have received any prescribed systemic or topical medication within 14 days of dosing with study drug unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety
3. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of dosing with study drug (with the exception of vitamin/mineral supplements and paracetamol) unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety
4. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of dosing with study drug unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety
5. Subjects who are still participating in a clinical study (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical or biological entity) in the past 3 months since the last dose.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
safety: adverse events | 13 days
  adverse events

SECONDARY OUTCOMES:
pharmacokinetics AUC | 13 days
  area under concentration time curve
pharmacokinetics Cmin | 13 days
  drug level in blood 24 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Frans van den Berg, MB ChB, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, UK, United Kingdom